CLINICAL TRIAL: NCT04743843
Title: Concordance Between Omnyx System With Omnyx .RTS Images and the Omnyx Dynamyx Software With Hamamatsu .NDPI Images
Status: Completed | Type: Observational
Sponsor: Inspirata Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-0042
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Omnyx Dynamyx Software — Digital pathology image management and viewing software.

SUMMARY:
This study serves as a validation study for the Omnyx Dynamyx software and Hamamatsu .ndpi image file format, evaluating agreement of diagnosis between whole slide images (WSI) of the Omnyx system (Omnyx scanned .rts images and Omnyx Dynamyx software) and the Omnyx Dynamyx software with the Hamamatsu .ndpi images. The primary goal of this study is to demonstrate concordance between the two systems to validate the Omnyx Dynamyx software with the non-Omnyx .ndpi image file type.

DETAILED DESCRIPTION:
The overall study design was to compare the diagnosis obtained by .rts WSI from the Omnyx system (Omnyx scanner and Omnyx Software) and diagnosis obtained by .ndpi WSI of the Hamamatsu S360 or similar scanner with the Omnyx Software. Pathologists read cases in the Omnyx Dynamyx software with .rts images from an Omnyx scanner and complete a Preliminary Surgical Pathology Consultant Report that includes a preliminary diagnosis. After a two-week washout period, the pathologists read the same cases in the Omnyx Dynamyx software with .ndpi images from a Hamamatsu scanner. The diagnosis from the Omnyx scanners are provided in the Final Surgical Pathology Consultant Report. Pathologists then complete an Inspirata Whole Slide Imaging Case Worksheet to determine confirmation of diagnosis - that is, agreement/concordance between the WSI from the two scanners.

The study is designed to prove that the diagnosis of a case will be the same when using the Omnyx .rts file type as the Hamamatsu .ndpi file type regardless of tissue or procedure type.

All discrepancies between the two "systems" will be documented and reconciled. Discrepancies categorized as Major or Minor. The Principal Investigator Discordance Review Form will be utilized to document the Principal Investigator's review of those cases where discrepancies were attributed to technical/technological aspects of WSI, such as sub-optimal image quality.

This is a deidentified, retrospective study to evaluate surgical pathology cases, excluding frozen sections and cytology. Formalin-fixed paraffin embedded tissue from sixty (60) cases across a range of three (3) subspecialist categories will be used.

Materials for each case include the original pathology report and the complete set of physical slides from each case at the time of diagnosis. Cases will be no more than two (2) years older than the Date of Protocol.

The pathology reports will be deidentified and the key to match the pathology reports with the deidentified physical slides and deidentified Whole Slide Images (WSI) will be retained and managed by the Study Sponsor.

Each slide will be scanned on the Omnyx VL120 scanner and Hamamatsu S360 scanner with 40x magnification settings and standard compression ratings for each system. Whole slide image data sets will be prepared by deidentified case number (for example, Case1- Case 60) and distributed to at least three (3) pathologists with any pertinent information about the case form the original pathology report EXCEPT the final diagnosis.

Each of the approximately 60 cases will be read in both the Omnyx system with Omnyx .rts images and the Omnyx Dynamyx software with Hamamatsu .ndpi images with a two (2) week wash-out period between the .rts and .ndpi case reads. Each case will only be read once (by the same pathologist) in each of the two modalities. Therefore, if three (3) pathologists participate, each pathologist will be responsible for reading twenty (20) cases in both image formats.

A pathologist will review all Omnyx .rts images first and record the preliminary diagnosis. The pathologist will then read the cases from the Hamamatsu .ndpi images in the Omnyx Dynamyx software and determine concordance between WSI produced by the Omnyx VL 120 scanner and viewed in the Omnyx Dynamyx software and images produced by the Hamamatsu S360 scanner and viewed in the Omnyx Dynamyx software. If the pathologist determines discordance, the PI will complete review of all discordant cases.

Concordance will be reported by subspecialty and overall and will be reported between the original pathology report and the .rts images and the .rts images and the .ndpi images. Discordance must be significant as discerned by the adjudication pathologist. Minor discordance will be measured but only significant discordance will be reported as a primary endpoint of this study.

ELIGIBILITY:
Inclusion Criteria:

* • Approximately 60 surgical pathology cases (20 from each sub-specialty group):

  * Dermatopathology;
  * Breast;
  * Head and Neck • Slides that are no more than 2 years old

Exclusion Criteria:

* • Frozen sections; and

  * Cytology cases
  * Slides that require special non-brightfield optical considerations such as polarization or fluorescence
  * Hematology slides
  * Slides that require 60x or higher magnification (oil immersion)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: • H&Es, IHCs and Special stains available at the time of the original diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Concordance between digitized .rts images and digitized .ndpi images | 3 months
  The proportion of diagnosis between Omnyx .rts images and Hamamatsu .ndpi images using Blyth-Still-Casella 95% confidence interval showed concordant diagnosis for each subspecialty and across all recommended subspecialties.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lloyd, Ph.D., Principal Investigator — Inspirata, Inc.
Locations (1):
- Northern Lincolnshire and Goole NHS Foundation Trust, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No